CLINICAL TRIAL: NCT03477084
Title: Understanding and Modelling Reservoirs, Vehicles and Transmission of ESBL-producing Enterobacteriaceae in the Community and Long Term Care Facilities
Brief Title: Understanding and Modeling Reservoirs, Vehicles and Transmission of ESBL-producing Enterobacteriaceae in the Community and Long Term Care Facilities
Acronym: MODERN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Hospital Universitario Virgen Macarena (Other); University Hospital Tuebingen (Other); University Hospital, Geneva (Other); UMC Utrecht (Other); University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: MODERN
Record Dates: First submitted 2018-03-12; First posted 2018-03-26 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2020-01

CONDITIONS: Resistance Bacterial; Enterobacteriaceae Infections
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample, environmental samples (wastewater, sinks, showers, food, toilets)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long Term Care Facilities: Spread of ESBL-producing E. coli and K. pneumoniae among the residents of Long Term Care Facilities.
  Interventions: Biological: ESBL-producing enterobacteriaceae carriage
- Households: Household transmission of ESBL-producing bacteria after hospital discharge of a patient carrying ESBL-producing E. coli or K. pneumoniae.
  Interventions: Biological: ESBL-producing enterobacteriaceae carriage

INTERVENTIONS:
Biological: ESBL-producing enterobacteriaceae carriage — Carriage of ESBL-producing Escherichia coli or Klebsiella pneumoniae

SUMMARY:
The continuing spread of extended-spectrum beta-lactamase-producing Enterobacteriaceae (ESBL-PE) is among the most important problems in antimicrobial resistance. It is also a good model to investigate the epidemiological complexity of resistance in Enterobacteriaceae. Available data on the transmission determinants of ESBL-PE in community settings are scarce, methodologically limited and mostly based on single centre studies. A comprehensive investigation using present typing and modelling techniques is warranted to develop a sound quantitative understanding of the interactions involved. A consortium of investigators with diverse expertise from countries with high and low endemicity of ESBL-EP has been created. Transmission and persistence of ESBL-PE within households and long-term care facilities will be studied. Individual and group-level determinants for transmission and persistence will be quantified, together with other ecological variables including environmental, food and wastewater contamination. Advanced molecular typing techniques and state of the art analytical methods will be used. Data generated in this project will directly inform a suite of mathematical models which, in addition to encapsulating current understanding of the processes, will be used to explore the potential effectiveness of different interventions to control ESBL-PE spread. The expected outputs are a comprehensive characterisation of ESBL-PE transmission considering bacterial clones and mobile genetic elements, as well as individual and ecologic-level factors in different settings, to inform public health authorities about interventions that should be prioritised to control transmission of these organisms.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the Bellevaux LTCF (Besançon - France)
* Patients discharged from the University Hospital of Besançon and carrying ESBL-E. coli or K. pneumoniae and their household members

Exclusion Criteria:

* Participation rejection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Residents of the Bellevaux LTCF (Besançon - France)
  * Patients discharged from the University Hospital of Besançon and carrying ESBL-E. coli or K. pneumoniae and their household members
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Transmission of ESBL-producing E. coli and K. pneumoniae (ESBL-E) in the community (LTCF residents and in households) | For the cohort 'LTCF': 35 weeks ; For the cohort 'Household': 4 months
  We will assess
  * For the cohort 'LTCF': the number of LTCF residents contaminated with an ESBL-E from other residents or from the environment within 35 weeks.
  * For the cohort 'Household': the number of people (sharing household with a ESBL-E carrying patient which has been discharged from the hospital) contaminated with ESBL-E within 4 months.
  These two measurements will be aggregated to arrive at one reported value : the number of secondary cases from one index case (ratio).

CONTACTS AND LOCATIONS:
Overall Officials: Elise Robert, Study Director — University Hospital of Besançon - France
Locations (1):
- University Hospital, Besançon, Bourgogne-Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No